CLINICAL TRIAL: NCT05386511
Title: An Observational, Real-world Study Study of UTD1 in Chinese Advanced Breast Cancer
Brief Title: Real-world Study of UTD1 in Chinese Advanced Breast Cancer
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Biyun Wang, MD, Professor, Fudan University
Other Study IDs: YOUNGBC-17
Record Dates: First submitted 2022-05-18; First posted 2022-05-23 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- UTD1: UTD1 monotherapy or UTD1 based therapy

SUMMARY:
To evaluate the efficacy and safety of UTD1 in patients with advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged over 18 years old.
2. Metastatic breast cancer included unresectable locally advanced breast cancer, de novo stage IV breast cancer, and recurrent metastatic breast cancer.
3. Plan to receive or has received UTD1 monotherapy or UTD1 based therapy
4. Available medical history.

Exclusion Criteria:

1.Incomplete medical history.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with breast cancer (according to ICD-10) with confirmed metastasis, regardless of being de novo diagnosed or progressed from a non-metastatic stage
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
PFS | 6 weeks
  Progression free survival

SECONDARY OUTCOMES:
Adverse events | 6 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided